CLINICAL TRIAL: NCT02703116
Title: Employing eSBI in a Community-based HIV Testing Environment for At-risk Youth
Brief Title: Employing eSBI in HIV Testing for At-risk Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Robert Garofalo, MD, Division Chief - Adolescent Medicine; Director - Center for Gender, Sexuality and HIV Prevention, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA041071 (NIH); R01DA041071 (NIH)
Record Dates: First submitted 2016-03-02; First posted 2016-03-09 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: HIV; Substance Use
Keywords: HIV; Substance Use
MeSH Terms: conditions — Substance-Related Disorders | interventions — Ethanol; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Use BI (Experimental): Those who are randomized to the intervention will complete eSBI, an electronic brief intervention for substance use, which is comprised of 11 topical areas, each with a single webpage, in a motivational interviewing (MI) format. MI is a client-centered behavioral change approach.
  Interventions: Behavioral: Alcohol Use BI
- Nutrition Intervention (Active Comparator): Those randomized to the control will complete the attention control modules, a non-active brief time-matched attention control intervention of equal length (i.e., encouraging nutrition).
  Interventions: Behavioral: Nutrition Intervention

INTERVENTIONS:
Behavioral: Alcohol Use BI — Those who are randomized to the intervention will complete eSBI, an electronic brief intervention for substance use, which is comprised of 11 topical areas, each with a single webpage, in a motivational interviewing (MI) format. MI is a client-centered behavioral change approach.
  Arms: Alcohol Use BI
Behavioral: Nutrition Intervention — Those randomized to the control will complete the attention control modules, a non-active brief time-matched attention control intervention of equal length (i.e., encouraging nutrition).
  Arms: Nutrition Intervention

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability and test the initial efficacy of eSBI, (electronic screening and brief intervention for alcohol use) coupled with STTR (Seek, Test, Treat, and Retain) in comparison to STTR only among YMSM (young men who have sex with men) and YTW (young transgender women) on frequency of substance use and engagement within the HIV (human immunodeficiency virus) and PrEP (pre-exposure prophylaxis) care continuum.

DETAILED DESCRIPTION:
The purpose of this study is to assess the feasibility, acceptability and test the initial efficacy of eSBI, (electronic screening and brief intervention for alcohol use) coupled with STTR (Seek, Test, Treat, and Retain) in comparison to STTR only among YMSM (young men who have sex with men) and YTW (young transgender women) on frequency of substance use and engagement within the HIV and PrEP (pre-exposure prophylaxis) care continuum. We will do this with the following aims:

Aim 1: Assess the feasibility, acceptability and initial efficacy of electronic Screening & Brief Intervention + Seek, Test, Treat and Retain (eSBI+ STTR) compared to STTR-only to reduce alcohol and other substance use among 450 YMSM and YTW in Chicago, ages 16-25, at 1, 3, 6, and 12 months post-intervention.

Aim 2: To explore the initial efficacy of eSBI+STTR in comparison to STTR-only on secondary exploratory outcomes within the HIV and PrEP care continuum among YMSM and YTW.

Aim 3: Determine the degree to which sub-groups of youth are differentially impacted by eSBI+STTR based on socio-demographic characteristics and co-morbid mental health problems to inform future targeting and/or tailoring of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged 16 to 25 years
* seeking testing for HIV infection
* HIV-negative or HIV status unknown (per self-report)
* Male who has had sex with men OR transgender woman who has had sex with men (i.e., born male, identify as female/transgender, and at any point in the gender transition process)
* English-speaking.

Exclusion Criteria:

* volunteer seems distraught or emotionally unstable (i.e. suicidal, manic, exhibiting violent behavior)
* volunteer seems intoxicated or under the influence of psychoactive agents

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male who has had sex with men OR transgender woman who has had sex with men (i.e., born male, identify as female/transgender, and at any point in the gender transition process)
Enrollment: 464 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Change in Frequency of Alcohol Use | 1, 3, 6 and 12 months post-intervention
  Self-reported frequency of alcohol use in the previous 1 and 12 months assessed via computer-assisted self-interviewing.

SECONDARY OUTCOMES:
PrEP and HIV-related Care Engagement | 1, 3, 6 and 12 months post-intervention
  PrEP and HIV-related medical care engagement (completed clinical visits) will be abstracted from medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Garofalo, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago; Niranjan Karnik, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (3):
- United States (3):
  - Ann & Robert H. Lurie Children's Hospital, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
Share de-identified study data upon request to study contacts and with approval from the principal investigator(s).
Time Frame: Post publication. Exact time frame undecided.
Access Criteria: Share de-identified study data upon request to study contacts and with approval from the principal investigator(s).

REFERENCES:
- [Derived] Karnik NS, Kuhns LM, Hotton AL, Del Vecchio N, McNulty M, Schneider J, Donenberg G, Keglovitz Baker K, Diskin R, Muldoon A, Rivera J, Summersett Williams F, Garofalo R. Findings From the Step Up, Test Up Study of an Electronic Screening and Brief Intervention for Alcohol Misuse in Adolescents and Young Adults Presenting for HIV Testing: Randomized Controlled Efficacy Trial. JMIR Ment Health. 2023 Mar 29;10:e43653. doi: 10.2196/43653. PMID 36989027
- [Derived] Kuhns LM, Karnik N, Hotton A, Muldoon A, Donenberg G, Keglovitz K, McNulty M, Schneider J, Summersett-Williams F, Garofalo R. A randomized controlled efficacy trial of an electronic screening and brief intervention for alcohol misuse in adolescents and young adults vulnerable to HIV infection: step up, test up study protocol. BMC Public Health. 2020 Jan 8;20(1):30. doi: 10.1186/s12889-020-8154-6. PMID 31914971